CLINICAL TRIAL: NCT01813227
Title: A Phase II Study of Carfilzomib in Relapsed Waldenström's Macroglobulinemia (WM) IST-CAR-531
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Onyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro 3596 (CAR-531)
Record Dates: First submitted 2013-03-11; First posted 2013-03-18 (Estimated); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — carfilzomib; Rituximab; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carfilzomib (Experimental): Carfilzomib 20 mg/m2 on day 1, 2 then 56 mg/m2 days 8, 9 and 15, 16 over 30 minutes every 28 days. Dexamethasone 4 mg (8 mg if > 45 mg/m2) orally each day of carfilzomib therapy. If less than a partial remission (PR) after 4 cycles, add rituximab 375 mg/m2 on day 16 of each cycle. Patients who meet the criteria for progression prior to 4 cycles of therapy will have rituximab added to their treatment. For patients receiving rituximab, the carfilzomib dose will be decreased to 27 mg/m2. Patients will be treated to maximal response plus 2 additional cycles to a maximum of 12 cycles.
  Interventions: Drug: Carfilzomib; Drug: Rituximab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — If you decide to participate in the study, you will receive carfilzomib on Days 1, 2, 8, 9, 15, and 16 every 28 days for a minimum of 2 cycles (approximately 2 months). You may receive additional cycles for as long as your disease remains stable or improved or until your study doctor determines that you should stop receiving the study drug or you decide to stop participating in the study.
  Other Names: Kyprolis
Drug: Rituximab — If you decide to participate in the study, in addition to the carfilzomib and possible dexamethasone administration, If less than a partial remission (PR) after 4 cycles is achieved, rituximab 375 mg/m2 on day 16 of each subsequent cycle will be added to the treatment. Subjects who meet the criteria for progression prior to 4 cycles of therapy will have rituximab 375 mg/m2 weekly for 4 consecutive weeks every 3 cycles added to the treatment. Subjects will be treated to maximal response plus 2 additional cycles to a maximum of 12 cycles.
  At the beginning of every cycle, your study doctor will see if your general health is satisfactory. You will be asked to report any side effects or problems you have had since the start of the last treatment cycle as well as any medication change(s).
  Other Names: Rituxan
Drug: Dexamethasone — If you decide to participate in the study, you will receive carfilzomib on Days 1, 2, 8, 9, 15, and 16 every 28 days for a minimum of 2 cycles (approximately 2 months). You may receive additional cycles for as long as your disease remains stable or improved or until your study doctor determines that you should stop receiving the study drug or you decide to stop participating in the study.
  You will also receive dexamethasone weekly on Days 1, 2, 8, 9, 15 and 16 starting with cycle 1 and continuing every cycle thereafter.
  Other Names: Decadron

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of an investigational study drug called carfilzomib. The investigators want to find out what effects, good and/or bad, it has on patients and their cancer if treatment continues beyond previous carfilzomib treatment study.

Carfilzomib (KyprolisTM) is approved by the U.S. Food and Drug Administration (FDA) to be used only in certain U.S. patients with relapsed and refractory multiple myeloma that have tried and failed other therapies. It has not been approved to be used for any other disease or condition.

In this study, carfilzomib is referred to as an investigational study drug because it is not approved for use in all patients with multiple myeloma in the United States, and it is not approved by some regulatory authorities (the agencies that are responsible for approving the use of a medicine in a country such as Health Canada).

Carfilzomib is a type of drug called a proteasome inhibitor. A proteasome is a protein found within cells that has the important role of identifying and marking damaged proteins that are needed to be destroyed by the cell for survival. The inhibition of the proteasome allows for damaged protein to accumulate within cells. This accumulation of damaged protein causes the cell to die.

DETAILED DESCRIPTION:
Waldenström's macroglobulinemia (WM) is a rare low-grade B-cell lymphoplasmacytic lymphoma. Overall reported incidences approximately 3 cases per million persons per year with about 1500 and cases diagnosed annually in United States. There is a higher incidence in males compared to females (3.4 vs 1.7 cases per 1 million person-years at risk) and WM is nearly twice as common among whites compared to blacks.[1] A familial form of the disease is also recognized. WM is an indolent disease with an overall median survival of 5 years although more recent data suggest a disease-specific median survival of 11.2 years, given the frequently older age (median 63 years) and accompanying co-morbidities at diagnosis(1). WM is characterized by infiltration of lymphoplasmacytic cells and bone marrow and by serum immunoglobulin M (IgM) monoclonal gammopathy. B-cell origin and some clinical cellular and epidemiological features are shared among WM arises from intermediately mature B cells (somatically mutated post germinal center the lymphocytes that have not yet undergone isotype switching), as opposed to immature B cells from which chronic lymphocytic leukemia arises in the fully mature, somatically mutated, from which cells multiple myeloma arises.

There is no standard of care for WM (2). Therefore, involving the patient's in clinical trials is strongly recommended whenever possible.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven WM with relapsed/refractory symptomatic disease are eligible for enrollment.
* Bone marrow lymphoplasmacytosis with:

  * > 10% lymphoplasmacytic cells (measured within 28 days prior to registration OR
  * Aggregates or sheets of one of the following: lymphocytes, plasma cells or lymphoplasmacytic cells on the bone marrow biopsy (measured within 28 days prior to registration).
  * Measurable disease defined as a quantitative IgM monoclonal protein of >500 mg/dL obtained within 28 days prior to registration
  * CD20+ bone marrow or lymph node by immunohistochemistry or flow cytometry obtained within 28 days prior to registration
  * Lymph node biopsy must be done <28 days prior to registration if used as an eligibility criterion for study entry.
* Symptomatic disease, as defined by the IWWM, includes the following criteria: Hemoglobin less than 10 g/dL, platelet count less than 100,000 uL, bulky adenopathy or organomegaly, symptomatic hyperviscosity syndrome, severe neuropathy, amyloidosis, cryoglobulinemia, cold agglutinin disease, or evidence of transformation high-grade non-Hodgkin's lymphoma.
* Patients must not be receiving concurrent steroids > 10 mg prednisone (or equivalent) per day.
* Prior irradiation is allowed if > 28 days prior to registration have elapsed since the date of last treatment.
* Women must not be pregnant or breast-feeding due to the fact that the reproductive risk to humans taking carfilzomib is unknown. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Women of childbearing potential and sexually active males must use an accepted and effective method of contraception throughout the study and for 8 weeks after completion of the study.
* Patients must be > 18 years old.
* Patients must have ECOG performance status of < 2.
* Patients may have received prior bortezomib therapy.
* Adequate hepatic function, with serum ALT ≤ 3times the upper limit of normal and serum direct bilirubin ≤ 2 mg/dL (34 µmol/L) within 14 days prior to randomization
* Absolute neutrophil count (ANC) ≥ 1.0 × 109/L within 14 days prior to randomization
* Hemoglobin ≥ 8 g/dL (80 g/L) within 14 days prior to randomization (subjects may be receiving red blood cell [RBC] transfusions in accordance with institutional guidelines)
* Platelet count ≥ 50 × 109/L (≥ 30 × 109/L if WM involvement in the bone marrow is > 50%) within 14 days prior to randomization
* Creatinine clearance (CrCl) ≥ 15 mL/minute within 7 days prior to randomization, either measured or calculated using a standard formula (e.g., Cockcroft and Gault)

Exclusion Criteria:

* Pre-existing peripheral neuropathy > grade 2 with pain (CTC version 4.0).
* Hematologic criteria: ANC < 500/uL, Platelets < 25,000 uL.
* Renal function: CrCl < 15 ml/min.
* Active infection requiring intravenous antibiotics
* Known Active hepatitis B or C
* SGOT (AST) and SGPT (ALT) > 3x institutional ULN
* Direct bilirubin > 1.5 mg/dL
* Patients must not have any severe and/or uncontrolled medical condition or other conditions that could affect their participation in the study, including, but not restricted to:
* Symptomatic congestive heart failure of New York Heart Association Class III or IV.
* Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 3 months of start of study treatment, serious uncontrolled cardiac arrhythmia or any other clinically significant heart disease.
* Severely impaired lung function as defined as spirometry and DLCO (corrected for Hgb) that is <50% of the normal predicted value and/or O2 saturation <88% at rest on room air.
* Active (acute or chronic) or uncontrolled severe infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Vesole, MD, PhD, Principal Investigator — John Theurer Cancer Center at Hackensack University Medical Center
Locations (1):
- John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Carfilzomib: Carfilzomib 20 mg/m2 on day 1, 2 then 56 mg/m2 days 8, 9 and 15, 16 over 30 minutes every 28 days. Dexamethasone 4 mg (8 mg if > 45 mg/m2) orally each day of carfilzomib therapy. If less than a partial remission (PR) after 4 cycles, add rituximab 375 mg/m2 on day 16 of each cycle. Patients who meet the criteria for progression prior to 4 cycles of therapy will have rituximab added to their treatment. For patients receiving rituximab, the carfilzomib dose will be decreased to 27 mg/m2. Patients will be treated to maximal response plus 2 additional cycles to a maximum of 12 cycles.
  Carfilzomib: Carfilzomib on Days 1, 2, 8, 9, 15, and 16 every 28 days for a minimum of 2 cycles (approximately 2 months). You may receive additional cycles for as long as your disease remains stable or improved or until your study doctor determines that you should stop receiving the study drug or you decide to stop participating in the study.
  Rituximab: If less than a partial remission (PR) after 4 cycles is achieved, rituximab 375 mg/m2 on day 16 of each subsequent cycle will be added to the treatment. Subjects who meet the criteria for progression prior to 4 cycles of therapy will have rituximab 375 mg/m2 weekly for 4 consecutive weeks every 3 cycles added to the treatment. Subjects will be treated to maximal response plus 2 additional cycles to a maximum of 12 cycles.
  Dexamethasone: weekly on Days 1, 2, 8, 9, 15 and 16 starting with cycle 1 and continuing every cycle thereafter.
Period: Overall Study
Arm/Group | Carfilzomib
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Carfilzomib
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 61.5 [56 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6
  African American | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) of Carfilzomib in Bortezomib naïve and Bortezomib-exposed Relapsed WM
Description: The overall response rate (ORR) (rate of patients attaining a Partial Response or a Complete Response). Responses will be based on both serum paraprotein levels by SPEP and bidimensional disease measurements on CT scan for patients with adenopathy/organomegaly/lymphadenopathy.
  Criteria as per the Recommended Response Criteria for Waldenstrom Macroglobulinemia
  Complete Response:
  * Absence of serum monoclonal IgM protein by immunofixation
  * Normal serum IgM level
  * Complete resolution of extramedullary disease, i.e., lymphadenopathy and splenomegaly if present at baseline
  * Morphologically normal bone marrow aspirate and trephine biopsy
  Partial response (PR)
  * Monoclonal IgM protein is detectable
    -≥50% but<90% reduction in serum IgM level from baseline
  * Reduction in extramedullary disease, i.e., lymphadenopathy/splenomegaly if present at baseline
  * No new signs or symptoms of active disease
Time Frame: Participants will be evaluated every 28 days (1 cycle) until progression or a maximum of 12 cycles (1 year)
Measure: Number; unit: percentage of participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 7
percentage of participants | 85.7

2. Secondary Outcome: Number of Patients Experiencing Dose Limiting Toxicity
Description: Number of Patients Experiencing Dose Limiting Toxicity.
Time Frame: Participants will be evaluated for the first 28 days of cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 7
Participants | 0

3. Secondary Outcome: Duration of Response in Patients With WM.
Time Frame: Participants will be evaluated every 28 days (1 cycle) until they experience disease progression, are treated with another therapy, or died, an average of 15 months
Measure: Mean (Full Range); unit: months
Arm/Group | Carfilzomib
Number analyzed (Participants) | 6
months | 15.4 [6.7 to 25.8]

4. Secondary Outcome: Time to Progression
Time Frame: Participants will be evaluated every 28 days (1 cycle) until disease progression, an average of 16 months
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Carfilzomib
Number analyzed (Participants) | 1
months | 16 (0)

5. Secondary Outcome: Progression Free Survival
Description: PFS will be censored at the last disease assessment visit for subjects who start alternative therapy or who are lost to follow up before documentation of disease progression or who are alive and do not have documentation of disease progression before a data analysis cutoff date
Time Frame: Participants will be evaluated every 28 days (1 cycle) until progression, an average of 19 months
Measure: Mean (Full Range); unit: months
Arm/Group | Carfilzomib
Number analyzed (Participants) | 7
months | 19.4 [12.7 to 26.7]

ADVERSE EVENTS:
Arm/Group | Carfilzomib
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib (N=7)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes